CLINICAL TRIAL: NCT03504280
Title: Changes in Serum Vitamin D Level and Clinical Parameters After Different Loading Doses of Cholecalciferol (D3) in Young Adults With Vitamin D Deficiency
Brief Title: Changes in Serum Vitamin D Level After Different Loading Doses of Cholecalciferol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr Shweta Nakarmi, Principle Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VitaminD
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Hypovitaminosis D
Keywords: hypovitaminosis D; cholecalciferol; mehadose
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: single center, interventional, open labelled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- high dose IM (Active Comparator): cholecalciferol 600,000 IU given intramuscularly
  Interventions: Drug: Cholecalciferol
- high dose oral (Active Comparator): cholecalciferol 600,000 IU given orally
  Interventions: Drug: Cholecalciferol
- low dose oral (Active Comparator): cholecalciferol 400,000 IU given orally in 2 divided doses given monthly for 2 consecutive months followed by daily maintenance dose of 1000 IU
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
it is a clinical trial to observe increase in serum vitamin D level and clinical symptoms after 3 different doses of cholecalciferol given either intramuscularly or oral.

DETAILED DESCRIPTION:
A prospective, interventional study was conducted in Department of Rheumatology, BSMMU, Dhaka, Bangladesh from October 2015 to January 2017. One hundred and five clinically healthy adults of age 21-39 with serum vitamin D concentration were enrolled in the study. Serum vitamin D level was estimated by chemiluminescent micro particle immunoassay method at baseline and 3 months after the intervention. The participants were divided into three groups using random number table. Group A was given 6 lakh IU of cholecalciferol IM stat dose, group B was given 6 lakh IU of cholecalciferol orally with a glass of milk stat dose and group c was given 2 lakh IU of cholecalciferol orally once a month for 2 months followed by tablet cholecalciferol 1000 IU daily.

ELIGIBILITY:
Inclusion Criteria:

* hypovitaminosis D (serum 25 OH D < 20 ng/ml)

Exclusion Criteria:

* Chronic disease causing Vitamin D deficiency like CKD, nephrotic syndrome, liver disease, hyperparathyroidism, history of skin graft, malabsorption, hyperthyroidism, drugs like anticonvulsants, glucocorticoids, HAART Current pregnancy Lactose intolerance Previously treated with bolus Vitamin D supplementation within previous three months

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D | 3 months
  serum vitamin D level in ng/ml measured by CLIA method

SECONDARY OUTCOMES:
fatigue | 3 months
  visual analog scale of fatigue during last 7 days of interview measured in 10 cm scale
generalized weakness | 3 months
  visual analog scale of generalized weakness during last 7 days of interview measured in 10 cm scale
bone pain | 3 months
  visual analog scale of bone pain during last 7 days of interview measured in 10 cm scale
muscle cramps | 3 months
  visual analog scale of muscle cramps during last 7 days of interview measured in 10 cm scale
pain in weight bearing joints | 3 months
  visual analog scale of pain in weight bearing joints during last 7 days of interview measured in 10 cm scale
difficulty in climbing stairs | 3 months
  visual analog scale of difficulty in climbing stairs during last 7 days of interview measured in 10 cm scale
difficulty in standing from squatting position | 3 months
  visual analog scale of difficulty in standing from squatting position during last 7 days of interview measured in 10 cm scale

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Nakarmi, resident, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Md Nazrul Islam, professor, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided